CLINICAL TRIAL: NCT00097734
Title: A Prospective, Multicenter, Open-Label, Randomized Clinical Study to Evaluate the Duration of Treatment With Ertapenem in Acute Attacks of Sigmoid Diverticulitis
Brief Title: Study to Evaluate the Duration of Treatment With Ertapenem in Acute Attacks of Sigmoid Diverticulitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum Hanover-Siloah Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: mc317; INVA-DIV-Study
Record Dates: First submitted 2004-11-29; First posted 2004-11-30 (Estimated); Last update posted 2006-02-14 (Estimated); Status verified 2006-02

CONDITIONS: Diverticulitis, Colonic; Acute Disease
Keywords: diverticulitis; Invanz; Ertapenem; acute attacks; sigmoid diverticulitis; Acute attacks of sigmoid diverticulitis
MeSH Terms: conditions — Diverticulitis, Colonic; Acute Disease; Diverticulitis | interventions — Ertapenem

INTERVENTIONS:
Drug: ertapenem

SUMMARY:
The purpose of this study is to compare the efficacy (by assessing the clinical success of treatment) of intravenous antibiotic therapy with ertapenem in patients with acute attacks of sigmoid diverticulitis for 4 vs. 7 days.

ELIGIBILITY:
Inclusion Criteria:

* At least three of the following signs or symptoms of an acute attack of sigmoid diverticulitis must be present: *Fever (body temperature > 38°C, sublingual), *Abdominal tenderness, *Leukocytosis (leukocytes > 10,000/µl) and left shift of the differential blood count (>1% band forms), *Elevated CRP (> 20 mg/l)
* Evidence of sigmoid diverticulitis by contrast enema
* CT evidence of wall thickening in the sigmoid intestine
* Decision in favor of conservative therapy on the basis of the case history and diagnosis

Exclusion Criteria:

* Contraindication for the use of the study medication or other beta-lactam antibiotics, e.g. patients with advanced renal impairment or patients requiring hemodialysis
* Antibiotic therapy in the two weeks prior to the start of the study
* Patients with an advanced incurable disease
* Patients with a hematologic/oncologic disease (leukemia, lymphoma)
* Patients on immunosuppressants
* Complications of sigmoid diverticulitis leading to an immediate indication for surgery
* Patients who have hypersensitivity to beta-lactam antibiotics
* Female patients who are pregnant or nursing or who could become pregnant during the study
* Participation in another clinical study or use of another study drug within the four weeks prior to enrollment in the study or use of another drug during the study
* Each patient can be enrolled only once in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2004-07; Study Completion 2007-06

PRIMARY OUTCOMES:
Clinical therapeutic success (full regression)
Relapse rate
Operation rate

SECONDARY OUTCOMES:
Development of laboratory parameters
Duration of hospitalization
Duration of parenteral feeding
Incidence of surgical intervention and repeat surgery
Incidence and duration of intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Koeckerling, Prof. Dr., Study Chair — Klinikum Hanover-Siloah hospital and Nordstadt hospital- Surgical Department
Locations (1):
- Klinikum Hannover- Krankenhaus Siloah, Hanover, Germany

REFERENCES:
- [Background] Ambrosetti P, Robert J, Witzig JA, Mirescu D, de Gautard R, Borst F, Meyer P, Rohner A. Prognostic factors from computed tomography in acute left colonic diverticulitis. Br J Surg. 1992 Feb;79(2):117-9. doi: 10.1002/bjs.1800790208. PMID 1555056
- [Background] Auguste L, Borrero E, Wise L. Surgical management of perforated colonic diverticulitis. Arch Surg. 1985 Apr;120(4):450-2. doi: 10.1001/archsurg.1985.01390280044010. PMID 3985790
- [Background] Bakker FC, Hoitsma HF, Den Otter G. The Hartmann procedure. Br J Surg. 1982 Oct;69(10):580-2. doi: 10.1002/bjs.1800691007. PMID 7127036
- [Background] Balthazar EJ, Robinson DL, Megibow AJ, Ranson JH. Acute pancreatitis: value of CT in establishing prognosis. Radiology. 1990 Feb;174(2):331-6. doi: 10.1148/radiology.174.2.2296641.
- [Background] Bell GA, Panton ON. Hartmann resection for perforated sigmoid diverticulitis. A retrospective study of the Vancouver General Hospital experience. Dis Colon Rectum. 1984 Apr;27(4):253-6. PMID 6714033
- [Background] Berry AR, Turner WH, Mortensen NJ, Kettlewell MG. Emergency surgery for complicated diverticular disease. A five-year experience. Dis Colon Rectum. 1989 Oct;32(10):849-54. doi: 10.1007/BF02554554. PMID 2791771
- [Background] BOLES RS Jr, JORDAN SM. The clinical significance of diverticulosis. Gastroenterology. 1958 Dec;35(6):579-82. No abstract available. PMID 13609810
- [Background] Chappuis CW, Cohn I Jr. Acute colonic diverticulitis. Surg Clin North Am. 1988 Apr;68(2):301-13. doi: 10.1016/s0039-6109(16)44479-8. PMID 3279548
- [Background] Cheskin LJ, Bohlman M, Schuster MM. Diverticular disease in the elderly. Gastroenterol Clin North Am. 1990 Jun;19(2):391-403. PMID 2194951
- [Background] Cheskin LJ, Lamport RD. Diverticular disease. Epidemiology and pharmacological treatment. Drugs Aging. 1995 Jan;6(1):55-63. doi: 10.2165/00002512-199506010-00005. PMID 7696779
- [Background] Cho KC, Morehouse HT, Alterman DD, Thornhill BA. Sigmoid diverticulitis: diagnostic role of CT--comparison with barium enema studies. Radiology. 1990 Jul;176(1):111-5. doi: 10.1148/radiology.176.1.2191360.
- [Background] Chodak GW, Rangel DM, Passaro E Jr. Colonic diverticulitis in patients under age 40: need for earlier diagnosis. Am J Surg. 1981 Jun;141(6):699-702. doi: 10.1016/0002-9610(81)90081-7. No abstract available. PMID 7246860
- [Background] Cunha BA. Ertapenem. A review of its microbiologic, pharmacokinetic and clinical aspects. Drugs Today (Barc). 2002 Mar;38(3):195-213. doi: 10.1358/dot.2002.38.3.820127. PMID 12532175
- [Background] Detry R, Jamez J, Kartheuser A, Zech F, Vanheuverzwijn R, Hoang P, Kestens PJ. Acute localized diverticulitis: optimum management requires accurate staging. Int J Colorectal Dis. 1992 Feb;7(1):38-42. doi: 10.1007/BF01647660. PMID 1588224
- [Background] Doringer E. Computerized tomography of colonic diverticulitis. Crit Rev Diagn Imaging. 1992;33(5):421-35. PMID 1418606
- [Background] Drusano GL, Warren JW, Saah AJ, Caplan ES, Tenney JH, Hansen S, Granados J, Standiford HC, Miller EH Jr. A prospective randomized controlled trial of cefoxitin versus clindamycin-aminoglycoside in mixed anaerobic-aerobic infections. Surg Gynecol Obstet. 1982 May;154(5):715-20. PMID 7041297
- [Background] Duma RJ, Kellum JM. Colonic diverticulitis: microbiologic, diagnostic, and therapeutic considerations. Curr Clin Top Infect Dis. 1991;11:218-47. No abstract available. PMID 1867769
- [Background] Eisenstat TE, Rubin RJ, Salvati EP. Surgical management of diverticulitis. The role of the Hartmann procedure. Dis Colon Rectum. 1983 Jul;26(7):429-32. doi: 10.1007/BF02556519. PMID 6861572
- [Background] Elsakr R, Johnson DA, Younes Z, Oldfield EC 3rd. Antimicrobial treatment of intra-abdominal infections. Dig Dis. 1998 Jan-Feb;16(1):47-60. doi: 10.1159/000016848. PMID 9549036
- [Background] Ertan A. Colonic diverticulitis. Recognizing and managing its presentations and complications. Postgrad Med. 1990 Sep 1;88(3):67-72; 77. doi: 10.1080/00325481.1990.11704725. PMID 2169049
- [Background] Eusebio EB, Eisenberg MM. Natural history of diverticular disease of the colon in young patients. Am J Surg. 1973 Mar;125(3):308-11. doi: 10.1016/0002-9610(73)90047-0. No abstract available. PMID 4690116
- [Background] Ferzoco LB, Raptopoulos V, Silen W. Acute diverticulitis. N Engl J Med. 1998 May 21;338(21):1521-6. doi: 10.1056/NEJM199805213382107. No abstract available. PMID 9593792
- [Background] Freischlag J, Bennion RS, Thompson JE Jr. Complications of diverticular disease of the colon in young people. Dis Colon Rectum. 1986 Oct;29(10):639-43. doi: 10.1007/BF02560326. PMID 3757703
- [Background] Barry AL, Fuchs PC, Brown SD. In vitro activity of the ketolide ABT-773. Antimicrob Agents Chemother. 2001 Oct;45(10):2922-4. doi: 10.1128/AAC.45.10.2922-2924.2001. PMID 11557491
- [Background] Goldstein EJ, Citron DM, Merriam CV, Warren Y, Tyrrell K. Comparative in vitro activities of GAR-936 against aerobic and anaerobic animal and human bite wound pathogens. Antimicrob Agents Chemother. 2000 Oct;44(10):2747-51. doi: 10.1128/AAC.44.10.2747-2751.2000. PMID 10991855
- [Background] Gottesman L, Zevon SJ, Brabbee GW, Dailey T, Wichern WA Jr. The use of water-soluble contrast enemas in the diagnosis of acute lower left quadrant peritonitis. Dis Colon Rectum. 1984 Feb;27(2):84-8. doi: 10.1007/BF02553980. PMID 6697835
- [Background] Hachigian MP, Honickman S, Eisenstat TE, Rubin RJ, Salvati EP. Computed tomography in the initial management of acute left-sided diverticulitis. Dis Colon Rectum. 1992 Dec;35(12):1123-9. doi: 10.1007/BF02251962. PMID 1473412
- [Background] Hackford AW, Schoetz DJ Jr, Coller JA, Veidenheimer MC. Surgical management of complicated diverticulitis. The Lahey Clinic experience, 1967 to 1982. Dis Colon Rectum. 1985 May;28(5):317-21. doi: 10.1007/BF02560431. PMID 3996147
- [Background] Haglund U, Hellberg R, Johnsen C, Hulten L. Complicated diverticular disease of the sigmoid colon. An analysis of short and long term outcome in 392 patients. Ann Chir Gynaecol. 1979;68(2):41-6. No abstract available. PMID 507737
- [Background] Hinchey EJ, Schaal PG, Richards GK. Treatment of perforated diverticular disease of the colon. Adv Surg. 1978;12:85-109. PMID 735943
- [Background] Hiltunen KM, Kolehmainen H, Vuorinen T, Matikainen M. Early water-soluble contrast enema in the diagnosis of acute colonic diverticulitis. Int J Colorectal Dis. 1991 Nov;6(4):190-2. doi: 10.1007/BF00341388. PMID 1770284
- [Background] HORNER JL. A study of diverticulitis of the colon in office practice. Gastroenterology. 1952 Jun;21(2):223-9. No abstract available. PMID 14937207
- [Background] Hulkko OA, Laitinen ST, Haukipuro KA, Stahlberg MJ, Juvonen TS, Kairaluoma MI. The Hartmann procedure for the treatment of colorectal emergencies. Acta Chir Scand. 1986 Aug-Sep;152:531-5. PMID 3788398
- [Background] Johnson CD, Baker ME, Rice RP, Silverman P, Thompson WM. Diagnosis of acute colonic diverticulitis: comparison of barium enema and CT. AJR Am J Roentgenol. 1987 Mar;148(3):541-6. doi: 10.2214/ajr.148.3.541. PMID 3492883
- [Background] Kellum JM, Sugerman HJ, Coppa GF, Way LR, Fine R, Herz B, Speck EL, Jackson D, Duma RJ. Randomized, prospective comparison of cefoxitin and gentamicin-clindamycin in the treatment of acute colonic diverticulitis. Clin Ther. 1992 May-Jun;14(3):376-84. PMID 1638578
- [Background] Kourtesis GJ, Williams RA, Wilson SE. Acute diverticulitis: safety and value of contrast studies in predicting need for operation. Aust N Z J Surg. 1988 Oct;58(10):801-4. doi: 10.1111/j.1445-2197.1988.tb00983.x. PMID 3250415
- [Background] Krukowski ZH, Matheson NA. Emergency surgery for diverticular disease complicated by generalized and faecal peritonitis: a review. Br J Surg. 1984 Dec;71(12):921-7. doi: 10.1002/bjs.1800711202. PMID 6388723
- [Background] Laitinen R, Tahtinen J, Lantto T, Vorne M. Tc-99m labeled leukocytes in imaging of patients with suspected acute abdominal inflammation. Clin Nucl Med. 1990 Sep;15(9):597-602. doi: 10.1097/00003072-199009000-00001. PMID 2208880
- [Background] Larson DM, Masters SS, Spiro HM. Medical and surgical therapy in diverticular disease: a comparative study. Gastroenterology. 1976 Nov;71(5):734-7. PMID 964566
- [Background] LEIGH JE, JUDD ES, WAUGH JM. Diverticulitis of the colon. Recurrence after apparently adequate segmental resection. Am J Surg. 1962 Jan;103:51-4. doi: 10.1016/0002-9610(62)90012-0. No abstract available. PMID 14463838
- [Background] Lindahl J, Ristkari SK, Vorne M, Mokka RE. 99m-technetium-HmPAO-labelled leucocytes in the diagnosis of acute colonic diverticulitis. Acta Chir Scand. 1989 Sep;155(9):479-82. PMID 2596257
- [Background] Ling L, Aberg T. Hartmann procedure. Acta Chir Scand. 1984;150(5):413-7. PMID 6435365
- [Background] Livermore DM, Carter MW, Bagel S, Wiedemann B, Baquero F, Loza E, Endtz HP, van Den Braak N, Fernandes CJ, Fernandes L, Frimodt-Moller N, Rasmussen LS, Giamarellou H, Giamarellos-Bourboulis E, Jarlier V, Nguyen J, Nord CE, Struelens MJ, Nonhoff C, Turnidge J, Bell J, Zbinden R, Pfister S, Mixson L, Shungu DL. In vitro activities of ertapenem (MK-0826) against recent clinical bacteria collected in Europe and Australia. Antimicrob Agents Chemother. 2001 Jun;45(6):1860-7. doi: 10.1128/AAC.45.6.1860-1867.2001. PMID 11353638
- [Background] Makela J, Vuolio S, Kiviniemi H, Laitinen S. Natural history of diverticular disease: when to operate? Dis Colon Rectum. 1998 Dec;41(12):1523-8. doi: 10.1007/BF02237300. PMID 9860333
- [Background] Mazuski JE, Sawyer RG, Nathens AB, DiPiro JT, Schein M, Kudsk KA, Yowler C; Therapeutic Agents Committee of the Surgical Infections Society. The Surgical Infection Society guidelines on antimicrobial therapy for intra-abdominal infections: evidence for the recommendations. Surg Infect (Larchmt). 2002 Fall;3(3):175-233. doi: 10.1089/109629602761624180. PMID 12542923
- [Background] McConnell EJ, Tessier DJ, Wolff BG. Population-based incidence of complicated diverticular disease of the sigmoid colon based on gender and age. Dis Colon Rectum. 2003 Aug;46(8):1110-4. doi: 10.1007/s10350-004-7288-4. PMID 12907908
- [Background] McGOWAN FJ, WOLFF WI. Diverticulitis of the sigmoid colon. Gastroenterology. 1952 May;21(1):119-32. No abstract available. PMID 14926820
- [Background] Morris J, Stellato TA, Lieberman J, Haaga JR. The utility of computed tomography in colonic diverticulitis. Ann Surg. 1986 Aug;204(2):128-32. doi: 10.1097/00000658-198608000-00005. PMID 3741003
- [Background] Murray JJ, Schoetz DJ Jr, Coller JA, Roberts PL, Veidenheimer MC. Intraoperative colonic lavage and primary anastomosis in nonelective colon resection. Dis Colon Rectum. 1991 Jul;34(7):527-31. doi: 10.1007/BF02049889. PMID 2055137
- [Background] Nagorney DM, Adson MA, Pemberton JH. Sigmoid diverticulitis with perforation and generalized peritonitis. Dis Colon Rectum. 1985 Feb;28(2):71-5. doi: 10.1007/BF02552645. PMID 3971809
- [Background] Nichols RL. Management of intra-abdominal sepsis. Am J Med. 1986 Jun 30;80(6B):204-9. doi: 10.1016/0002-9343(86)90502-4. PMID 3524217
- [Background] Odenholt I, Lowdin E, Cars O. In vitro pharmacodynamic studies of L-749,345 in comparison with imipenem and ceftriaxone against gram-positive and gram-negative bacteria. Antimicrob Agents Chemother. 1998 Sep;42(9):2365-70. doi: 10.1128/AAC.42.9.2365. PMID 9736564
- [Background] Painter NS. Diverticular disease of the colon. The first of the Western diseases shown to be due to a deficiency of dietary fibre. S Afr Med J. 1982 Jun 26;61(26):1016-20. PMID 6283684
- [Background] Papi C, Ciaco A, Koch M, Capurso L. Efficacy of rifaximin in the treatment of symptomatic diverticular disease of the colon. A multicentre double-blind placebo-controlled trial. Aliment Pharmacol Ther. 1995 Feb;9(1):33-9. doi: 10.1111/j.1365-2036.1995.tb00348.x. PMID 7766741
- [Background] Parks TG. Natural history of diverticular disease of the colon. A review of 521 cases. Br Med J. 1969 Dec 13;4(5684):639-42. doi: 10.1136/bmj.4.5684.639. PMID 5359917
- [Background] Parks TG, Connell AM. The outcome in 455 patients admitted for treatment of diverticular disease of the colon. Br J Surg. 1970 Oct;57(10):775-8. doi: 10.1002/bjs.1800571021. No abstract available. PMID 5476757
- [Background] Perkins JD, Shield CF 3rd, Chang FC, Farha GJ. Acute diverticulitis. Comparison of treatment in immunocompromised and nonimmunocompromised patients. Am J Surg. 1984 Dec;148(6):745-8. doi: 10.1016/0002-9610(84)90429-x. PMID 6507744
- [Background] Pontari MA, McMillen MA, Garvey RH, Ballantyne GH. Diagnosis and treatment of enterovesical fistulae. Am Surg. 1992 Apr;58(4):258-63. PMID 1586086
- [Background] Porta E, Germano A, Ferrieri A, Koch M. The natural history of diverticular disease of the colon: a role for antibiotics in preventing complications? A retrospective study. Riv Eur Sci Med Farmacol. 1994 Jan-Apr;16(1-2):33-9. PMID 7761680
- [Background] Rege RV, Nahrwold DL. Diverticular disease. Curr Probl Surg. 1989 Mar;26(3):133-89. doi: 10.1016/0011-3840(89)90031-2. PMID 2651018
- [Background] Roberts P, Abel M, Rosen L, Cirocco W, Fleshman J, Leff E, Levien D, Pritchard T, Wexner S, Hicks T, et al. Practice parameters for sigmoid diverticulitis. The Standards Task Force American Society of Colon and Rectal Surgeons. Dis Colon Rectum. 1995 Feb;38(2):125-32. doi: 10.1007/BF02052438. PMID 7851165
- [Background] Sarin S, Boulos PB. Evaluation of current surgical management of acute inflammatory diverticular disease. Ann R Coll Surg Engl. 1991 Sep;73(5):278-82. PMID 1929127
- [Background] Shah PM, Isaacs RD. Ertapenem, the first of a new group of carbapenems. J Antimicrob Chemother. 2003 Oct;52(4):538-42. doi: 10.1093/jac/dkg404. Epub 2003 Sep 1. No abstract available. PMID 12951340
- [Background] Smith TR, Cho KC, Morehouse HT, Kratka PS. Comparison of computed tomography and contrast enema evaluation of diverticulitis. Dis Colon Rectum. 1990 Jan;33(1):1-6. doi: 10.1007/BF02053191. PMID 2295271
- [Background] Solomkin JS, Yellin AE, Rotstein OD, Christou NV, Dellinger EP, Tellado JM, Malafaia O, Fernandez A, Choe KA, Carides A, Satishchandran V, Teppler H; Protocol 017 Study Group. Ertapenem versus piperacillin/tazobactam in the treatment of complicated intraabdominal infections: results of a double-blind, randomized comparative phase III trial. Ann Surg. 2003 Feb;237(2):235-45. doi: 10.1097/01.SLA.0000048551.32606.73. PMID 12560782
- [Background] Schechter S, Mulvey J, Eisenstat TE. Management of uncomplicated acute diverticulitis: results of a survey. Dis Colon Rectum. 1999 Apr;42(4):470-5; discussion 475-6. doi: 10.1007/BF02234169. PMID 10215046
- [Background] Schwerk WB, Schwarz S, Rothmund M. Sonography in acute colonic diverticulitis. A prospective study. Dis Colon Rectum. 1992 Nov;35(11):1077-84. doi: 10.1007/BF02252999. PMID 1425053
- [Background] Starnes HF Jr, Lazarus JM, Vineyard G. Surgery for diverticulitis in renal failure. Dis Colon Rectum. 1985 Nov;28(11):827-31. doi: 10.1007/BF02555486. PMID 3902414
- [Background] Taylor KJ, Wasson JF, De Graaff C, Rosenfield AT, Andriole VT. Accuracy of grey-scale ultrasound diagnosis of abdominal and pelvic abscesses in 220 patients. Lancet. 1978 Jan 14;1(8055):83-4. doi: 10.1016/s0140-6736(78)90016-8. PMID 74578
- [Background] Tellado J, Woods GL, Gesser R, McCarroll K, Teppler H. Ertapenem versus piperacillin-tazobactam for treatment of mixed anaerobic complicated intra-abdominal, complicated skin and skin structure, and acute pelvic infections. Surg Infect (Larchmt). 2002 Winter;3(4):303-14. doi: 10.1089/109629602762539535. PMID 12697078
- [Background] Thompson WG, Patel DG. Clinical picture of diverticular disease of the colon. Clin Gastroenterol. 1986 Oct;15(4):903-16. PMID 3536213
- [Background] Tyau ES, Prystowsky JB, Joehl RJ, Nahrwold DL. Acute diverticulitis. A complicated problem in the immunocompromised patient. Arch Surg. 1991 Jul;126(7):855-8; discussion 858-9. doi: 10.1001/archsurg.1991.01410310065009. PMID 1854245
- [Background] Ulin AW, Pearce AE, Weinstein SF. Diverticular disease of the colon: surgical perspectives in the past decade. Dis Colon Rectum. 1981 May-Jun;24(4):276-81. doi: 10.1007/BF02641877. PMID 6972290
- [Background] Verbanck J, Lambrecht S, Rutgeerts L, Ghillebert G, Buyse T, Naesens M, Tytgat H. Can sonography diagnose acute colonic diverticulitis in patients with acute intestinal inflammation? A prospective study. J Clin Ultrasound. 1989 Nov-Dec;17(9):661-6. doi: 10.1002/jcu.1870170909. PMID 2514202
- [Background] WAUGH JM, WALT AJ. Current trends in the surgical treatment of diverticulitis of the sigmoid colon. Surg Clin North Am. 1962 Oct;42:1267-76. doi: 10.1016/s0039-6109(16)36792-5. No abstract available. PMID 13999257
- [Background] Wexner SD, Dailey TH. The initial management of left lower quadrant peritonitis. Dis Colon Rectum. 1986 Oct;29(10):635-8. doi: 10.1007/BF02560324. PMID 3757702
- [Background] Woods RJ, Lavery IC, Fazio VW, Jagelman DG, Weakley FL. Internal fistulas in diverticular disease. Dis Colon Rectum. 1988 Aug;31(8):591-6. doi: 10.1007/BF02556792. PMID 3402284
- [Background] WELCH CE, ALLEN AW, DONALDSON GA. An appraisal of resection of the colon for diverticulitis of the sigmoid. Ann Surg. 1953 Sep;138(3):332-43. doi: 10.1097/00000658-195313830-00005. No abstract available. PMID 13080959